CLINICAL TRIAL: NCT03801811
Title: Prospective Observational Study on the Safety and Efficacy of Cyanoacrylate Skin Glues to Reduce the Risk of Complications After Insertion of Totally Implantable Central Venous Catheters Port-a-Cath
Brief Title: Use of the Skin Glue in the Placement of Central Venous Catheters Port a Catch
Acronym: Port glue cvc
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Parma (Other)
Responsible Party: Principal Investigator, Elena Giovanna Bignami, Professor, University of Parma
Other Study IDs: 382/2018/DISP/AOUPR
Record Dates: First submitted 2018-12-28; First posted 2019-01-14 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2018-09

CONDITIONS: Central Venous Catheter
Keywords: Port; Glue; CVC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Study of the efficacy of using skin glue in the application of Port a cath — The use of glue as a device in the implantation of central venous catheters has recently been introduced into European clinical practice. It is possible that the surgical incision created for the insertion of the PORT may be subject to complications such as: local bleeding, which if not properly treated may last even a few days, infections or surgical wound outbreaks. This possibility of bleeding occurs more easily in patients suffering from coagulation problems or when appropriate preventive measures have not been taken at the time of implantation of the device. A solution to this problem could be the application of the cyanoacrylate dermal glue on the edges of the surgical wound, after intradermal suture. The glue would have the purpose of sealing the surgical wound so as to immediately seal the skin incision with hemostatic effect and create a potential barrier against bacterial infections.

SUMMARY:
The use of glue as a device in the implantation of central venous catheters has recently been introduced into European clinical practice, initially with the aim of blocking bleeding at the point of exit of the PICCs, but at the same time also to close the cutaneous incision practiced to create the PORT positioning pocket.

It is possible that the surgical incision created for the insertion of the PORT may undergo complications such as: local bleeding, infections or wounds of the surgical wound.

A solution to this problem could be the application of the cyanoacrylate dermal glue on the edges of the surgical wound, after intradermal suture. The glue would have the purpose of sealing the surgical wound so as to immediately seal the skin incision with hemostatic effect and create a potential barrier against infections.

DETAILED DESCRIPTION:
Patient's informed consent signature for adhesion at the study will be initially requested. With their acceptance, parameters will be recorded anonymously in the Case Report Form, identified by a numeric code, until hospital discharge.

The parameters analized will be related to:

* essential patient data (identification number, gender, age, height weight)
* basic diseases
* associated diseases and risk factors
* origin of the patient (department or home)
* reason for positioning
* hemorrhagic complications detected in the first 24 hours
* hemorrhagic complications detected in the first 7 days
* non-bleeding complications detected at 7 days (local and systemic infections, wound delescence)

The data wil be transferred to an Excel worksheet, in order to conduct a descriptive analysis related to every variable

ELIGIBILITY:
Inclusion Criteria:

* informed consent signature
* age > 18 years

Exclusion Criteria:

* Age> 90 years
* Cianoacrilate allergy
* Presence of bacteraemia
* Informed consent refusal

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: critical ill patients
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-09-05 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
visible presence of blood around the emergency site | 24 hours
  Evaluate the effectiveness of cyanoacrylate glue in reducing / eliminating bleeding local from the insertion site after PORT implantation (evaluated as visible presence of blood around the emergency site.

SECONDARY OUTCOMES:
Early infection of the emergency site; | 7 days
  Rate of early infection of the emergency site; Early infection of the emergency site is assessed by observing skin changes as the presence of: pain, hot skin and reddened skin
Deischence of the surgical wound | 15 days
  Rate of dehiscence of the surgical wound. This will be assessed by looking for signs of bleeding, pain, fever and inflammation
Systemic infection | 15 days
  Rate of systemic infections will be evaluated by evaluating the presence of fever

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Universitaria di Parma, Parma, Italy